CLINICAL TRIAL: NCT06402643
Title: Comparative Analysis of Recurrence Rate Between Mini-Slet (Simple Limbal Epithelial Transplantation) Versus Limbal-Conjunctival Autograft Techniques in Primary Pterygium Excision
Brief Title: Comparison of Recurrence Between Mini-SLET and Limbal-Conjunctival Autograft Techniques in Primary Pterygium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, Enrique Graue, Head of the Cornea and Refractive Surgery Department, Instituto de Oftalmología Fundación Conde de Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI-049-2023
Record Dates: First submitted 2024-04-15; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pterygium of Right Eye; Pterygium of Left Eye; Pterygium of Both Eyes; Pterygium
Keywords: Pterygium,; Mini-SLET; Conjunctival-Limbal autograft
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Intervention Model Description: The allocation sequence will be generated by an investigator and will
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The allocation of the study participants will be concealed in opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-SLET. (Experimental): In addition to the standard resection technique, the surgical procedure will include the application of AM with surgical adhesive at the surgical site. Following this, limbal cells will be harvested from the limbus in a resection measuring 2×2 mm, divided into six fragments, and positioned along the limbus border on the AM.
  Interventions: Procedure: Pterygium Excision
- Conjunctival-Limbal Autograft. (Active Comparator): Pterygium will be surgically removed utilizing conventional resection techniques, entailing a blunt resection of the head, neck, and body of the pterygium. Subsequent to the resection, the surgical site will be polished using a surgical diamond burr if deemed necessary, and hemostasis will be achieved using bipolar cautery. In the case of CLAu, an autograft will be procured from the superior temporal bulbar conjunctiva. The autograft will be fixed to the surgical site using surgical adhesive.
  Interventions: Procedure: Pterygium Excision

INTERVENTIONS:
Procedure: Pterygium Excision — Pterygium will be surgically removed utilizing conventional resection techniques, entailing a blunt resection of the head, neck, and body of the pterygium. Subsequent to the resection, the surgical site will be polished using a surgical diamond burr if deemed necessary, and hemostasis will be achieved using bipolar cautery.

SUMMARY:
The surgical treatment options for pterygium, an abnormal growth on the eye's frontal surface can be treated with several surgical techniques. The rates of pterygium coming back varies depending on the surgical technique employed and other factors related to the patient and surgery. The objective of this study is to assess the efficacy and safety of incorporating a single amniotic membrane with stem cells in the treatment of primary pterygium, aiming to enhance surgical outcomes and minimize recurrence rates.

DETAILED DESCRIPTION:
The surgical treatment options for pterygium, an abnormal growth on the eye's surface, encompass various approaches. These include standard surgical excision, which involves removing the pterygium using traditional surgical methods and more recently Simple Limbal Epithelial Transplantation. Recurrence rate of pterygium varies depending on the surgical technique employed and other factors related to the patient and surgery.The objective of this study is to assess the efficacy and safety of incorporating a single amniotic membrane with stem cells in the treatment of primary pterygium, aiming to enhance surgical outcomes and minimize recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary nasal pterygium > 2mm
* Patients who can present and continue follow-up for the duration of the study
* Acceptance to participate in the study by signing the informed consent.

Exclusion Criteria:

* Patients with rheumatoid arthritis
* Collagenopathy
* Pregnant
* Infection, conjunctival inflammation or ocular trauma
* Glaucoma
* Previous ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-06-22 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1 month, 3, months, 6 months and 12 months after surgery.
  Any fibrovascular growth that passes onto the cornea across the limbus, will be considered a recurrence.

SECONDARY OUTCOMES:
Postoperative symptoms | 1 month, 3, months, 6 months and 12 months after surgery.
  Any postoperative symptoms, such as: pain, foreign body sensation, irritation, and tearing.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de oftalmología conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vera-Duarte GR, Ortiz-Morales G, Muller-Morales CA, Navas A, Ramirez-Miranda A, Graue-Hernandez EO, Kahuam-Lopez N. Mini-simple limbal epithelial transplantation and conjunctival-limbal autograft for the treatment of primary pterygium: Study protocol for a randomized controlled trial. Trials. 2025 Oct 31;26(1):457. doi: 10.1186/s13063-025-09075-3. PMID 41174752